CLINICAL TRIAL: NCT00856570
Title: An Open-label, One-sequence Crossover Study to Evaluate the Effect of Multiple Doses of YM178 on the Pharmacokinetics of Warfarin in Healthy Subjects
Brief Title: A Clinical Study to Determine the Effect of YM178 on the Pharmacokinetics of Warfarin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-040; EudraCT 2008-000211-15
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Overactive Bladder; Pharmacokinetics
Keywords: YM178; Mirabegron; DDI; Phase I; Warfarin; Pharmacokinetics
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Warfarin; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: warfarin — Oral
  Other Names: Coumadin
Drug: YM178 — Oral
  Other Names: mirabegron

SUMMARY:
This study investigates whether YM178 has an effect on the pharmacokinetics of warfarin, to exclude any drug-drug interaction between YM178 and warfarin, and evaluates the safety and tolerability of warfarin alone and combined with YM178.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must be of non-child bearing potential, i.e. postmenopausal, surgically sterilized (e.g. tubal ligation), hysterectomy in medical history, or must practice adequate (double barrier) non-hormonal contraceptive methods to prevent pregnancies.
* Body Mass Index (BMI) ≥ 18.5 and < 30 kg/m2, inclusive

Exclusion Criteria:

* Female who is pregnant
* Any of the liver function tests (i.e. alanine aminotransferase (ALT), aspartate aminotransferase (AST) and Alkaline Phosphatase (AP)) above the upper limit of normal (ULN)
* Any clinically significant history of disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Abnormal pulse and/or blood pressure measurements and the pre-study as follows: Pulse < 40 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (blood measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically
* A marked baseline prolongation of QT/QTc interval after repeated measurements of >450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* Use of any prescribed or OTC (over-the counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for paracetamol (up to 3 g/day)
* Any use of drugs of abuse within 3 months prior to admission to the clinical unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit
* History of drinking more than 21 units of alcohol per week (1 unit = 270 ml of beer or 40 ml of spirits or 1 glass of wine) (> 14 units of alcohol for female subjects) within 3 months prior to admission to the clinical unit
* Donation of blood or blood products within 3 months prior to admission to the clinical unit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
R- and S-warfarin in plasma: AUCinf, AUClast, Cmax, tmax, t1/2, CL/F | Day 1-9 and 15-31
The AUCinf of both enantiomers will be used to assess the potential drug-drug interaction. | Day 1/2 and 15/16

SECONDARY OUTCOMES:
Adverse events, clinical laboratory tests (hematology, biochemistry, urinalysis), vital signs, 12-lead ECG, physical examination | Day -1 - 31
YM178 in plasma: Ctrough, AUCtau, Cmax, tmax, CL/F | Day 20-24
Degree of anticoagulation: AUCPT;0-168h (area under the prothrombin time versus time curve from 0 to 168 h after dosing with warfarin), AUCINR;0-168h, maximum PT (PTmax), time to reach PTmax (tPT; max), INRmax, tINR;max | Day 1-9 and 23-31

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Paris, France